CLINICAL TRIAL: NCT04119986
Title: Safety and Efficacy of Drug Coated Balloon Therapy for Coronary In-stent Restenosis in Patients With Coronary Heart Disease Under the Guidance of QFR (UNIQUE-DCB-II Study)
Brief Title: Safety and Efficacy of DCB Therapy for ISR Under the Guidance of QFR (UNIQUE-DCB-II Study )
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY201910
Record Dates: First submitted 2019-10-07; First posted 2019-10-09 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Coronary Heart Disease
Keywords: Quantitative flow ratio; drug coated balloon; Drug eluted stent; In-stent restenosis
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- drug coated balloon (Experimental): A total of 110 patients with ISR are assigned to drug coated balloon treated group after randomization schedule.
  Interventions: Device: drug coated balloon
- drug eluted stent implantation (Other): A total of 110 patients with ISR are assigned to drug eluted stent treated group after randomization schedule.
  Interventions: Device: drug eluted stent

INTERVENTIONS:
Device: drug coated balloon — Balloon/vessel diameter ratio 0.8-1.0, 8-12 ATM (atmosphere), lasting for >30 seconds.
  Arms: drug coated balloon
Device: drug eluted stent — with regular techniques
  Arms: drug eluted stent implantation

SUMMARY:
In 1970, the first percutaneous balloon coronary angioplasty opened a new chapter of interventional therapy. However, the incidence of intracoronary restenosis was about 30%. Subsequently, bare metal stents and drug-eluting stents (DES) reduced the incidence of in-stent restenosis (ISR) to 5%-10% and it was still a bottleneck treated by percutaneous coronary intervention (PCI). Currently, ISR is mainly treated by balloon angioplasty, stent implantation and coronary artery bypass grafting.

In 2014, the guidelines of the European Society of Cardiology recommended that drug balloon therapy (DCB) and new generation DES should be the preferred strategies for ISR treatment. Compared with DES, DCB treatment can avoid the inflammation of intima caused by multi-layer stent strut, and reduce the risk of intimal hyperplasia and thrombosis in stent. However, DCB lacks sustained radial support. Even if the residual stenosis is less than 30% after sufficient pre-dilation, the elastic retraction of the intima still exists. In addition, the antiproliferative effect of paclitaxel is significantly worse than that of sirolimus and its derivatives, and there is a lack of long-term sustained release of anti-proliferative drugs. Compared with DCB, DES can obtain long-term stable radial support and long-term anti-proliferation effect, but stent struts exposed in the vascular lumen are at risk of stent thrombosis. The new generation of DES improves the design of stent platform, improves the polymer coating, and applies new anti-proliferative drugs. It effectively reduces the inflammation of vascular wall, speeds up the process of vascular re-endothelialization, promotes early vascular repair, and significantly reduces the incidence of stent thrombosis. Recent BIOLUXRCT, RESTORE and DARE studies provide more powerful evidence for the treatment of ISR by new generation DES.

Quantitative flow ratio (QFR) is the second generation FFR detectional method based on coronary contrast image. The latest FAVOR II results also confirm that QFR is more sensitive and specific than quantitative coronary analysis (QCA) in the diagnosis of myocardial ischemia caused by coronary artery stenosis. However, there is no report of ISR treated with DCB under the guidance of QFR. The aim of this study was to evaluate the safety and efficacy of DCB in the treatment of in-stent restenosis in patients with coronary heart disease (CHD) under the guidance of QFR compared with DES implantation.

DETAILED DESCRIPTION:
The current study is designed as a multicenter, randomized and prospective study aiming to evaluate the safety and efficacy of drug balloon therapy for ISR in patients with CHD under the guidance of QFR compared with DES implantation. Based on previous study reported, the incidence rate of target lesion failure is about 3% in patients with ISR undergoing DES implantation. And the design of non-inferiority study was performed in our study. Moreover, the investigators estimated 10% loss follow-up of these patients in each arm. As a result, a total of 220 patients with ISR were required, and with 110 patients per group as a ratio of 1:1 randomization.

ELIGIBILITY:
Inclusion Criteria:

● Meet the diagnostic criteria for patients with coronary in-stent restenosis and QFR<0.8 of target lesion in the coronary stent

Exclusion Criteria:

* QFR less than 0.8, dissection above type B and thrombosis formation after pre-dilation of ISR
* Severe congestive heart failure [LVEF <30% or NYHA( New York Heart Association) III/IV)]
* Severe valvular heart disease
* Life expectancy no more than 1 year or factors causing difficulties in clinical follow up
* Intolerance to aspirin and/or clopidogrel
* Known intolerance or allergy to heparin, contrast agents, paclitaxel, iopromide, rapamycin, polylactic acid-glycolic acid copolymer, Co-Cr alloy or platinum-chromium alloy
* Leukopenia or thrombopenia
* A history of peptic ulcer or GI bleeding in the previously
* Stroke within 6 months prior to the operation
* A history of severe hepatic or renal failure

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
The incidence rate of late lumen loss after percutaneous coronary intervention in patients with ISR | Follow-up coronary angiography at 12 months after the procedure
  The incidence rate of late lumen loss between DCB treated group and DES treated group evaluated by quantitative coronary analysis in patients with ISR

SECONDARY OUTCOMES:
The incidence rate of patient-related ischemic events | Clinical follow up at 30 days, 6, 9 and 12 months after the operation
  The incidence rate of patient-related ischemic events including all myocardial infarction, any revascularization and all-cause death

CONTACTS AND LOCATIONS:
Overall Officials: Fei Ye, MD, Principal Investigator — Nanjing First Hospital, Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kolh P, Windecker S, Alfonso F, Collet JP, Cremer J, Falk V, Filippatos G, Hamm C, Head SJ, Juni P, Kappetein AP, Kastrati A, Knuuti J, Landmesser U, Laufer G, Neumann FJ, Richter DJ, Schauerte P, Sousa Uva M, Stefanini GG, Taggart DP, Torracca L, Valgimigli M, Wijns W, Witkowski A; European Society of Cardiology Committee for Practice Guidelines; Zamorano JL, Achenbach S, Baumgartner H, Bax JJ, Bueno H, Dean V, Deaton C, Erol C, Fagard R, Ferrari R, Hasdai D, Hoes AW, Kirchhof P, Knuuti J, Kolh P, Lancellotti P, Linhart A, Nihoyannopoulos P, Piepoli MF, Ponikowski P, Sirnes PA, Tamargo JL, Tendera M, Torbicki A, Wijns W, Windecker S; EACTS Clinical Guidelines Committee; Sousa Uva M, Achenbach S, Pepper J, Anyanwu A, Badimon L, Bauersachs J, Baumbach A, Beygui F, Bonaros N, De Carlo M, Deaton C, Dobrev D, Dunning J, Eeckhout E, Gielen S, Hasdai D, Kirchhof P, Luckraz H, Mahrholdt H, Montalescot G, Paparella D, Rastan AJ, Sanmartin M, Sergeant P, Silber S, Tamargo J, ten Berg J, Thiele H, van Geuns RJ, Wagner HO, Wassmann S, Wendler O, Zamorano JL; Task Force on Myocardial Revascularization of the European Society of Cardiology and the European Association for Cardio-Thoracic Surgery; European Association of Percutaneous Cardiovascular Interventions. 2014 ESC/EACTS Guidelines on myocardial revascularization: the Task Force on Myocardial Revascularization of the European Society of Cardiology (ESC) and the European Association for Cardio-Thoracic Surgery (EACTS). Developed with the special contribution of the European Association of Percutaneous Cardiovascular Interventions (EAPCI). Eur J Cardiothorac Surg. 2014 Oct;46(4):517-92. doi: 10.1093/ejcts/ezu366. Epub 2014 Aug 29. No abstract available. PMID 25173601
- [Background] Wong YTA, Kang DY, Lee JB, Rha SW, Hong YJ, Shin ES, Her SH, Nam CW, Chung WY, Kim MH, Lee CH, Lee PH, Ahn JM, Kang SJ, Lee SW, Kim YH, Lee CW, Park SW, Park DW, Park SJ. Comparison of drug-eluting stents and drug-coated balloon for the treatment of drug-eluting coronary stent restenosis: A randomized RESTORE trial. Am Heart J. 2018 Mar;197:35-42. doi: 10.1016/j.ahj.2017.11.008. Epub 2017 Nov 22. PMID 29447782
- [Background] Xu B, Tu S, Qiao S, Qu X, Chen Y, Yang J, Guo L, Sun Z, Li Z, Tian F, Fang W, Chen J, Li W, Guan C, Holm NR, Wijns W, Hu S. Diagnostic Accuracy of Angiography-Based Quantitative Flow Ratio Measurements for Online Assessment of Coronary Stenosis. J Am Coll Cardiol. 2017 Dec 26;70(25):3077-3087. doi: 10.1016/j.jacc.2017.10.035. Epub 2017 Oct 31. PMID 29101020